CLINICAL TRIAL: NCT04043260
Title: Evaluation of the DreaMed Advisor Pro System in Subjects With Type 1 Diabetes Treated With Multiple Daily Injections of Insulin
Brief Title: DreaMed Advisor Pro System in Subjects With Type 1 Diabetes Treated With MDI Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DreaMed Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-0998
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Insulin-dependent Diabetes Mellitus; Diabetes Mellitus, Type 1
Keywords: Diabetes Type 1; Multiple Daily Injections
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Subject's glucose and insulin data will be transferred to the DreaMed Advisor Pro system. Optimization of insulin treatment plan will be done using the DreaMed Advisor Pro algorithm. After approval by the study physician (may override the suggestions for safety reasons), the treatment plan will be sent to the subject to be followed for the following 3 weeks. The study team will follow-up with a phone call to the subject to verify the subject received the updated treatment plan.
  Interventions: Device: Advisor Pro

INTERVENTIONS:
Device: Advisor Pro — The DreaMed Advisor Pro software is a proprietary algorithm, designed to provide a comprehensive analysis of individual diabetes data which consists of glucose levels and insulin delivery history. the Advisor Pro algorithm identifies glucose patterns and their possible causes, which may hamper the patient's glucose control, and recommend on adjustment to the patient-specific insulin treatment profiles as well as suggestions for personalized diabetes management tips (such as timing of meal boluses, bolus delivery compliance and personalized glucose targets).

SUMMARY:
A multi center, open label, prospective study that will include up to 100 subjects with Type 1 Diabetes treated with Multiple Daily Injections (MDI) of insulin according to a predefined sliding scale plan or carbohydrate ratio (CR) and correction factor (CF) plan, and Self-Monitoring of Blood Glucose (SMBG) or Continuous Glucose Monitoring (CGM).

The study will include screening, a 3-4 weeks run-in period and a 6 weeks intervention period. Subjects will be asked to record their insulin delivery during basal/bolus insulin treatment (using dedicated apps and/or connected pens) and their daily activities (meals, physical activity etc.) using electronic log (implemented on Dedicated Apps), for a total period of 9-10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Documented T1D for at least 1 year prior to study enrolment
2. Subjects aged 18 - 65 years old
3. A1c at inclusion ≤ 10%
4. Subjects using basal-bolus MDI therapy:

   1. Basal insulin: Glargine, Degludec, or Determir
   2. Bolus insulin: regular insulin, rapid analogues or ultra-rapid analogues
5. Subjects using CGM or SMBG that are compatible with data transmission to the study DMS.
6. BMI < 28 kg/m2
7. Subjects willing to follow study instructions:

   1. For SMBG users: measure capillary blood glucose at least 4 times a day and twice a week 7-point profile (optional). Document blood glucose level, insulin delivery, meals and daily activities. Wear blinded CGM.
   2. For CGM users: Use CGM according to manufacture instructions, Document insulin delivery, meals and daily activities.
8. Subjects have connection to the internet at home.
9. Subjects have a smartphone compatible with study requirements
10. Subjects willing and able to sign a written informed consent form.

Exclusion Criteria:

1. An episode of diabetic keto-acidosis within the month prior to study entry and/or severe hypoglycemia resulting in seizure or loss of consciousness in the month prior to enrolment.
2. Concomitant diseases/ treatment that influence metabolic control or any significant diseases /conditions including psychiatric disorders and substance abuse that in the opinion of the investigator is likely to affect the subject's ability to complete the study or compromise patients' safety
3. Relevant severe organ disorders (diabetic nephropathy, diabetic retinopathy, diabetic foot syndrome) or any secondary disease or complication of diabetes mellitus, such as:

   * Subject has unstable or rapidly progressive renal disease or is receiving dialysis
   * Subject has active proliferative retinopathy
   * Active gastroparesis
4. Participation in any other interventional study
5. Female subject who is pregnant or planning to become pregnant within the planned study duration
6. Subject is in the "honeymoon" phase - i.e. less than 0.5 insulin units/kg per day.
7. Drug or alcohol abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Percentage of readings below 54 mg/dl | 9 weeks
  Compare percentage of readings below 54 mg/dl during 3 weeks run-in period to percentage of readings below 54 mg/dl during intervention period.

SECONDARY OUTCOMES:
Percentage of readings within range of 70-180 mg/dl | 9 weeks
Change in HbA1C post study treatment | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yael Shtrit, Study Director — DreaMed Diabetes Ltd.
Locations (1):
- Schneider MC, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No